CLINICAL TRIAL: NCT03018301
Title: Effect of Single Intravenous Ketamine Dose on Postoperative Pain Following Cesarean Section Under Spinal Anesthesia: A Randomized Control Clinical Trial.
Brief Title: Intravenous Ketamine and Postoperative Pain Following Cesarean Section.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrady S Ibrahim, MD, Assistant professor of anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB0000871238
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine group (Active Comparator): will receive 0.25 mg/kg intravenous ketamine diluted with normal saline to 20 ml delivered over 10 minutes.
  Interventions: Drug: Ketamine
- Control group (Placebo Comparator): will receive intravenous 20 ml of normal saline, delivered over 10 minutes.
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Ketamine — will receive 0.25 mg/kg intravenous ketamine diluted with normal saline to 20 ml delivered over 10 minutes.
  Other Names: Ketalar
  Arms: Ketamine group
Other: Normal saline — will receive intravenous 20 ml of normal saline, delivered over 10 minutes.
  Arms: Control group

SUMMARY:
The purpose of this study is to investigate the analgesic effect of low-dose intravenous ketamine in pregnant mothers undergoing cesarean section under Bupivacaine spinal anesthesia.

DETAILED DESCRIPTION:
* No premedication will be given, and patients will be monitored by electrocardiogram, non-invasive arterial blood pressure, and pulse oximetry when they entered the operating room.
* 18 gauge IV cannula will be inserted and all patients will be preloaded with 10 ml/kg of lactate ringer over 20 min period.
* All participants will have spinal anesthesia using bupivacaine. The dose of the drug, as well as the method of injection will be identical for all individuals; 10 mg (2 cc 0.5%), in the L4-L5 space using needle 25 G, midline, with the patient in a sitting position.
* After administering bupivacaine, and prior to surgery the height of the sensory block will be assessed bilaterally (complete loss of sensation to ice) in a ascending fashion starting from T12 dermatome.
* Once adequate anesthesia to at least T6 dermatome will be achieved, the operation will be allowed to begin. When systolic blood pressure decrease to < 90 mmHg, or 30% of the pre-anesthetic blood pressure, it will be corrected by administering 5 mg ephedrine.
* Patients will be asked to report any intraoperative pain using visual pain score(VPS)of 0(no pain) 10(worst pain).

ELIGIBILITY:
Inclusion Criteria:

* Eligible women ASA class 1 and 2, are at term (≥37 week gestation), Scheduled for elective cesarean section whose anesthetic plan is for spinal anesthesia with Bupivacaine and intravenous pethidine and paracetamol for post operative analgesia.

Exclusion Criteria:

* • Body mass index ≥40 kg/m2,

  * Known allergy to any of the study medications,
  * Contraindication to the spinal anesthesia,
  * History of substance abuse,
  * History of hallucinations,
  * Chronic opioid therapy,
  * Chronic pain.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
• Number of Subjects Requiring Supplemental Analgesia | 24 hours postoperative

SECONDARY OUTCOMES:
Cumulative morphine/paracetamol | 24 hours postoperative
Number of subjects reporting nausea, vomiting | 24 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Israa M Sayed, Study Chair — Assiut University
Locations (1):
- Assiut university faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] El-Tahan MR, Warda OM, Yasseen AM, Attallah MM, Matter MK. A randomized study of the effects of preoperative ketorolac on general anaesthesia for caesarean section. Int J Obstet Anesth. 2007 Jul;16(3):214-20. doi: 10.1016/j.ijoa.2007.01.012. Epub 2007 Apr 24. PMID 17459695